CLINICAL TRIAL: NCT03108885
Title: Measuring Cell Free DNA During the Course of Treatment for Esophageal Cancer as a Marker of Response and Recurrence
Status: Terminated | Type: Observational
Why Stopped: Study's Principal Investigator no longer at the institution.
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 16-010506
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Neoplasm; Esophageal Neoplasms Malignancy Unspecified; Esophageal Neoplasms Malignant; Cancer of Esophagus; Cancer of the Esophagus; Esophageal Cancer; Esophagus Cancer; Neoplasm, Esophageal
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Blood Specimen Collection; Tissue Banks

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will have blood drawn prior to any neoadjuvant treatment or surgery. Tumor tissue will be collected and stored after pathologic evaluation has been completed. Blood collections will then be drawn at every subsequent follow up visit at Mayo Clinic for surveillance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood and Tissue Collection — Blood DNA will be isolated from plasma. Tumor DNA will be purified with a kit and amplified regions of 10 genes discovered to by mutated in whole exome sequencing.

SUMMARY:
To prospectively collect blood and tumor tissue from esophageal cancer patients to identify specific esophageal cancer mutations that can be measured in the blood (cell free DNA) during the course of treatment as a marker of response and recurrence.

DETAILED DESCRIPTION:
Esophageal carcinoma is an aggressive malignancy and about a third of patients present with distant metastatic disease. While survival is slowly improving with better diagnostic tools and therapy, the overall 5-year survival remains low at 18%. Unlike other malignancies, such as colon cancer and prostate cancer, there is no peripheral blood marker of response or recurrence during treatment in esophageal cancer. However, quantifying cfDNA is a unique and tumor specific avenue that may allow real time response to treatment in esophageal cancer.

To identify esophageal cancer specific mutations, tumor samples will undergo whole exome sequencing. From this data, the investigators will select 10-15 genes to focus their efforts. PCR primers will be designed to detect these tumor specific mutations in the cell-free component of peripheral blood samples over the course of treatment for esophageal cancer.

The investigators will obtain baseline blood (before treatment) and then collect blood after neoadjuvant treatment, after surgery, and then at subsequent visits from the participants.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal Cancer any stage
* Age >18 years old
* Willing and able to provide consent
* No prior history of neoadjuvant therapy for the esophageal cancer

Exclusion Criteria:

* Age <18 years old
* Unable to provide consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Undergoing surgery and follow up at Mayo Clinic Rochester for esophageal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Esophageal Cancer Mutation | 5 years
  To identify specific esophageal cancer mutations that can be measured in the blood (cell free DNA) during the course of treatment as a marker of response and recurrence.

SECONDARY OUTCOMES:
Marker for Recurrence | 5 years
  To validate cfDNA as a marker of recurrence of esophageal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Shanda Blackmon, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials